CLINICAL TRIAL: NCT07245433
Title: Evaluating the Effect of Xylitol Wipes on Cariogenic Bacteria in Infants and Toddlers: A Longitudinal Clinical Trial
Brief Title: Evaluating the Effect of Xylitol Wipes on Cariogenic Bacteria in Infants and Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Omar Abdelsadek, BDS, MSc, PhD, Professor of Pediatric Dentistry, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Faculty of Dentistry
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Early Childhood Caries (ECC); Dental Caries Prevention; Oral Bacterial Colonization; Pediatric Oral Health
Keywords: xylitol wipes; mutans streptococci; lactic acid; early childhood caries; clinical trial

STUDY DESIGN:
Intervention Model Description: Single-group, before-after longitudinal design. All enrolled children (9 months to 1.5 years) received the same intervention: mothers used commercially available xylitol dental wipes for their child 3 times daily for 4 weeks (4.2g/day). Outcomes (salivary lactic acid via Clinpro Cario-L-Pop and mutans streptococci counts via CRT kit) were measured at baseline and weekly for 4 visits. Compliance and adverse events were checked at each visit. No randomization or masking.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Xylitol Wipe Intervention (Experimental): All participants (children aged 9-18 months) in this single-arm study received the same intervention. Mothers were instructed to use commercially available xylitol dental wipes to clean their child's teeth and gums three times daily after meals for four weeks. Each wipe provided an estimated total daily xylitol exposure of about 4.2 g.
  The purpose of the intervention was to evaluate its preventive effect on early childhood caries by reducing cariogenic bacterial activity. The primary outcomes measured were:
  Salivary lactic acid levels using the Clinpro Cario-L-Pop chairside test kit. Mutans streptococci counts using the CRT bacteria caries risk test. All children were monitored weekly for compliance, oral health status, and any minor side effects. No comparator or placebo arm was included.
  Interventions: Other: Xylitol Dental Wipes

INTERVENTIONS:
Other: Xylitol Dental Wipes — Commercially available xylitol dental wipes were used for daily oral cleaning in infants and toddlers. Mothers were instructed to wipe their child's teeth and gums three times daily after meals for four consecutive weeks. Each wipe contained a xylitol-based solution providing a total daily exposure of approximately 4.2 g of xylitol. The intervention aimed to reduce cariogenic bacterial activity and prevent early childhood caries. Compliance, tolerance, and any minor side effects were recorded weekly during follow-up visits.

SUMMARY:
This clinical study evaluates whether cleaning infants' and toddlers' teeth and gums with xylitol-containing wipes can help reduce oral bacteria associated with early childhood caries. A total of 20 healthy children aged 9 to 18 months are enrolled. Mothers are instructed to clean their children's teeth and gums using xylitol dental wipes three times daily after meals for four weeks. Saliva samples are collected at baseline and during weekly follow-up visits to measure lactic acid levels and mutans streptococci counts. A pediatric dentist examines each child at every visit to monitor general oral health and to check for any potential side effects. The study aims to assess the feasibility, safety, and potential preventive value of parent-applied xylitol wipes during early childhood.

DETAILED DESCRIPTION:
This longitudinal interventional study is designed to assess the preventive effect of xylitol-containing dental wipes on oral bacteria linked to early childhood caries (ECC). The study enrolls 20 healthy, caries-free infants and toddlers aged 9 to 18 months attending the Pediatric Dentistry Department, Faculty of Dentistry, Alexandria University. After obtaining informed consent, mothers are instructed to use commercially available xylitol dental wipes (Spiffies Baby Tooth Wipes™, Dr. Products Inc., USA) to clean their children's teeth and gums three times daily after meals for four consecutive weeks. Each wipe contains a xylitol-based solution intended to provide mechanical cleaning and daily exposure to approximately 4.2 g of xylitol.

Saliva samples are collected at baseline and at four weekly follow-up visits. Two primary outcome measures are assessed:

Lactic acid levels, using the Clinpro Cario-L-Pop chairside kit (3M ESPE, Germany) Mutans streptococci counts, using the CRT Bacteria Caries Risk Test (Ivoclar Vivadent, Liechtenstein) Participants are monitored weekly to assess compliance, document any dietary changes, and report potential side effects, including mild gastrointestinal symptoms. Children undergo oral examinations by a pediatric dentist at each visit to evaluate oral tissues and overall tolerance of the intervention.

The study protocol focuses on determining whether the regular use of xylitol wipes is feasible, acceptable to parents and children, and potentially useful as a preventive measure against early childhood oral bacterial activity.

ELIGIBILITY:
Inclusion Criteria:

Healthy infants and toddlers aged 9 months to 18 months

Caries-free (no visible dental decay or white spot lesions)

Cooperative child and mother willing to participate for 4 weeks

Mother able to understand and follow instructions for xylitol wipe use

Written informed consent obtained from parent or legal guardian

Exclusion Criteria:

Infants or toddlers with systemic diseases or medical conditions affecting saliva

Use of antibiotics or antimicrobial mouth products within the past 4 weeks

Known allergy or sensitivity to xylitol or product components

Existing oral lesions or ongoing dental treatment

Non-compliance with study protocol or loss to follow-up

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Change in salivary lactic acid level | Baseline; weeks 1, 2, 3, and 4.
  Description: Lactic acid level in saliva measured using the Clinpro Cario-L-Pop chairside kit.
  Unit of Measure: Lactic acid score (1-9 scale).
Change in salivary mutans streptococci (MS) count | Baseline; weeks 1, 2, 3, and 4.
  Description: Mutans streptococci colony density assessed using the CRT bacteria caries risk test.
  Unit of Measure: MS score (0-3 scale).

SECONDARY OUTCOMES:
Parental compliance and tolerance to xylitol wipes | Weekly for 4 weeks.
  Description: Compliance is assessed by the number of wipes used per day, as reported by mothers during weekly interviews. During the same visits, mothers are asked whether any minor side effects (such as gastrointestinal discomfort or irritation) occurred in the child; these observations are recorded for monitoring purposes but are not treated as separate outcome variables.
  Unit of Measure: Number of wipes used per day.

OTHER OUTCOMES:
Ease of xylitol wipe application | Weekly for 4 weeks.
  Description: Ease of application is assessed weekly using a structured questionnaire in which mothers rate how easy or difficult it was to use the xylitol wipes. During these interviews, mothers also report the child's acceptance of the wipe application (e.g., acceptance or refusal) and provide general feedback on satisfaction and willingness to continue use. These observations are recorded for context but are not treated as separate outcome variables.
  Unit of Measure: Ease-of-use rating (easy / moderate / difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Omar A El Meligy, BDS,MSc,PhD, Principal Investigator — Alexandria University; Laila M El-Habashy, BDS,MSc,PhD, Principal Investigator — Alexandria University and Pharos University; Aliaa A Hamouda, BDS,MSc,PhD, Study Chair — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not or might not be shared due to the small sample size and privacy concerns involving infant participants.

REFERENCES:
- [Result] Babu V, Hegde S, Bhat S, Sargod S. Evaluation of Efficacy of Three Different Commercially Available Kit for Chairside Cariogenic Bacteria Test - Caries Risk Test, Saliva-check Mutans and CariScreen. Cureus. 2019 Dec 29;11(12):e6504. doi: 10.7759/cureus.6504. PMID 32025425
- [Result] Galganny-Almeida A, Queiroz MC, Leite AJ. The effectiveness of a novel infant tooth wipe in high caries-risk babies 8 to15 months old. Pediatr Dent. 2007 Jul-Aug;29(4):337-42. PMID 17867402
- [Result] Soderling E, Pienihakkinen K. Specific effects of xylitol chewing gum on mutans streptococci levels, plaque accumulation and caries occurrence: a systematic review. BMC Oral Health. 2025 Jul 29;25(1):1275. doi: 10.1186/s12903-025-06602-1. PMID 40731400
- [Result] Soderling EM. Xylitol, mutans streptococci, and dental plaque. Adv Dent Res. 2009;21(1):74-8. doi: 10.1177/0895937409335642. No abstract available. PMID 19717413
- [Result] Miyasawa-Hori H, Aizawa S, Takahashi N. Difference in the xylitol sensitivity of acid production among Streptococcus mutans strains and the biochemical mechanism. Oral Microbiol Immunol. 2006 Aug;21(4):201-5. doi: 10.1111/j.1399-302X.2006.00273.x. PMID 16842502
- [Result] Kishi M, Abe A, Kishi K, Ohara-Nemoto Y, Kimura S, Yonemitsu M. Relationship of quantitative salivary levels of Streptococcus mutans and S. sobrinus in mothers to caries status and colonization of mutans streptococci in plaque in their 2.5-year-old children. Community Dent Oral Epidemiol. 2009 Jun;37(3):241-9. doi: 10.1111/j.1600-0528.2009.00472.x. PMID 19508271